CLINICAL TRIAL: NCT04281862
Title: DEXTENZA Compared to Topical Prednisolone in Patients Undergoing Bilateral LASIK
Brief Title: DEXTENZA Compared to Topical Prednisolone in Patients Undergoing Bilateral LASIK Surgery
Acronym: AtLAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ATLAS2020
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Refractive Surgery
MeSH Terms: interventions — Calcium Dobesilate; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Dextenza
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Group B (Active Comparator): Topical Prednisolone
  Interventions: Drug: Topical Prednisolone

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — The insert, containing 0.4 mg of active pharmaceutical product, is placed within the canaliculus to provide a sustained and tapered delivery of drug to the ocular surface over 30 days after a one-time insertion. The attributes of the insert reduce the risks for improper corticosteroid tapering and unwanted peaks and troughs in drug concentration.
  Arms: Group A
Drug: Topical Prednisolone — Standard of care topical drop treatment
  Arms: Group B

SUMMARY:
To determine patient preference and treatment outcomes with an intracanalicular dexamethasone (0.4mg) insert compared to standard steroid drop regimen in the contralateral eye following bilateral LASIK surgery.

DETAILED DESCRIPTION:
This prospective, open-label, single-center, randomized, investigator-sponsored clinical study seeks to investigate the outcomes of patients undergoing bilateral LASIK surgery with the treatment of a dexamethasone intracanalicular insert compared to standard of care topical prednisolone. All eyes will receive treatment. Additionally, all eyes will receive topical moxifloxacin QID for 1 week.

Twenty patient eyes undergoing bilateral LASIK surgery will be randomized to receive either Dextenza (Group A) OR standard of care prednisolone acetate 1% QID for 1 week, BID for 1 week (Group B). The contralateral eye will receive treatment with either DEXTENZA or topical prednisolone as a comparator based on randomization of first eye to Group A or Group B. Post-operative evaluations will be performed on Day 1, Day 7, and Month 1 following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient who is planned to undergo bilateral LASIK surgery.
* Refractive error between the 2 eyes of 2 Diopters or less
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Patients under the age of 18.
* Patients who choose to have monovision after LASIK
* Patients with corneal pathology that may interfere with LASIK outcomes
* Patients who are pregnant (must be ruled out in women of child-bearing age with pregnancy test).
* Active infectious ocular or systemic disease.
* Patients with active infectious ocular or extraocular disease.
* Patients actively treated with local or systemic immunosuppression including systemic corticosteroids.
* Patients with known hypersensitivity to Dexamethasone.
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator.
* Patients with a history of ocular inflammation or macular edema.
* Patients with allergy or inability to receive topical antibiotic.
* Patients on systemic non-steroidal anti-inflammatory drugs (NSAID) greater than 1,200 mg/day
* Patients with a corticosteroid implant (i.e. Ozurdex).
* Active or history of chronic or recurrent inflammatory eye disease in either eye
* Ocular pain in either eye
* Proliferative diabetic retinopathy in either eye
* Significant macular pathology detected on macular optical coherence tomography evaluation at the screening visit in either eye
* Laser or incisional ocular surgery during the study period and 6 months prior in either eye
* History of cauterization of the punctum

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Patient Preference | Through Month 1 (Day 28 +/- 3 days)
  As measured by COMTOL adapted survey.
Patient Comfort | Through Month 1 (Day 28 +/- 3 days)
  As measured by SPEED Questionnaire.

SECONDARY OUTCOMES:
Ocular Surface Health | Through Month 1 (Day 28 +/- 3 days)
  As measured by corneal staining.
Visual Outcomes | Through Month 1 (Day 28 +/- 3 days)
  As measured by uncorrected Visual Acuity.
Ocular Pain | Through Month 1 (Day 28 +/- 3 days)
  As measured by Ocular Pain Assessment.

OTHER OUTCOMES:
Safety Endpoints | Through Month 1 (Day 28 +/- 3 days)
  As measured by intraocular pressure increase of 10 mm Hg or greater from baseline.
Safety Endpoints | Through Month 1 (Day 28 +/- 3 days)
  As measured by proportion of eyes rescued with additional topical prednisolone treatment or increased frequency of dosing.
Safety Endpoints | Through Month 1 (Day 28 +/- 3 days)
  As measured by occurrence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Vance Thompson Vision ND, West Fargo, North Dakota, United States